CLINICAL TRIAL: NCT00006441
Title: A Single Center, Randomized Open Label Study of Initial Interleukin-2 Compared to Delayed Interleukin-2 When Added to Zidovudine, 3TC and Nelfinavir In Order to Modulate Immune Function and to Sustain Suppression of HIV-1 Replication Among Those Persons With Primary or Early HIV Infection
Brief Title: Effectiveness of Adding Interleukin-2 to Anti-HIV Drugs in Patients Recently Infected With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Chiron Corporation (Industry); Agouron Pharmaceuticals (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI-01-001; AIEDRP AI-01-001; 10435 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2000-11-03; First posted 2001-08-31 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: Virus Replication; HIV-1; Interleukin-2; Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; CD4-Positive T-Lymphocytes; CD8-Positive T-Lymphocytes; Biological Markers; Lamivudine; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Nelfinavir; Cytotoxicity, Immunologic; Acute Infection
MeSH Terms: conditions — HIV Infections | interventions — lamivudine, zidovudine drug combination; Nelfinavir; aldesleukin; Interleukin-2

ARMS (2):
- A (Experimental): Patients beginning IL-2 treatment regimens after 4 weeks of study
  Interventions: Drug: Lamivudine/Zidovudine; Drug: Nelfinavir mesylate; Drug: Aldesleukin
- B (Active Comparator): Patients beginning IL-2 treatment after some delay based on specified criteria
  Interventions: Drug: Lamivudine/Zidovudine; Drug: Nelfinavir mesylate; Drug: Aldesleukin

INTERVENTIONS:
Drug: Lamivudine/Zidovudine — 300/150 mg respectively twice daily for 104 weeks. Patients who develop intolerence to AZT may use Stavudine (d4T) at a dose of 40 mg daily.
  Other Names: Combivir
Drug: Nelfinavir mesylate — 1250 mg twice daily for 104 weeks.
  Other Names: NFV
Drug: Aldesleukin — 7.5 million units twice daily. Treatment will last until conclusion of study.
  Other Names: IL-2

SUMMARY:
The purpose of this study is to see whether taking interleukin-2 (IL-2) and other anti-HIV drugs affects the course of HIV disease in patients with primary HIV infection (the time period that immediately follows infection with HIV).

After primary HIV infection, the actual infection is spread through an increasing amount of HIV virus in the body. Studies have shown that, by taking a combination of anti-HIV drugs, it is possible to reduce the amount of HIV in the body to almost undetectable levels. This study will find out if starting anti-HIV drugs during primary infection will interrupt or reduce the spread of HIV in patients' bodies.

DETAILED DESCRIPTION:
Following initial exposure to HIV, infection is established through the rapid replication of a homogeneous strain of the virus. Preliminary studies of combination antiretroviral therapy show that it is possible to reduce circulating HIV RNA to below detectable levels at this phase. Sustained suppression of viral replication or viral eradication may be possible only before HIV has become integrated in the immune system and undergone a number of quasi species mutations. This study will assess the feasibility of interrupting the natural course of HIV infection by using antiretroviral therapy soon after initial infection.

Nelfinavir (NFV) and zidovudine/lamivudine (Combivir) treatment starts as soon as possible and at most, 7 days from the diagnosis of HIV infection, and continues for 104 weeks. After 4 weeks of therapy patients are randomized to begin receiving IL-2 therapy or to delay starting it until Week 48. Patients may choose not to receive IL-2 treatment and remain in the study. Patients have clinic visits to measure viral load every 4 weeks. At a final clinic visit, physical examinations and collection of semen, cervical fluid, blood, and saliva specimens are done. Eligible consenting patients have a tonsil biopsy. Patients are reimbursed for participation in this study.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Have recent HIV infection.
* Are available for follow-up for at least 96 weeks.
* Are at least 18 years old.
* Use a barrier method of birth control.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a condition such as Epstein-Barr virus, CMV mononucleosis syndrome, or acute streptococcal pharyngitis.
* Have taken anti-HIV therapy for over 4 weeks.
* Have or have had cancer requiring chemotherapy or radiation therapy within 1 month of study entry and have not yet recovered from the effects.
* Abuse alcohol and other drugs.
* Are pregnant.
* Have a condition which interferes with intestinal absorption, such as severe diarrhea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2003-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the dynamics of HIV in different tissue compartments of maximally suppressive antiretroviral (ART) medications with IL-2 influences, viral pathogenesis and immune responses to HIV infection. | Throughout study
To determine the patterns of immunologic activation as measured by cell surface marker levels, soluble and cell-associated cytokines when persons with acute or early HIV infection are treated with ART and IL-2. | Throughout study
To examine whether the extent of CD8+ cell antiviral activity as measured by non-cytotoxic and cytotoxic responses affects the kinetics of viral replication and viral load in blood plasma. | Throughout study
To determine whether a broad cellular immune response to HIV infection, measured by T cell repertoire, cytotoxic T cell lymphocyte function and CD4 T helper function correlates with the patterns of cellular immune antiviral responses | Throughout study

SECONDARY OUTCOMES:
To follow a cohort of HIV negative individuals that tested with the Options Project to use as a comparison group with the HIV positive individuals enrolling in this protocol. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Jay Levy, Principal Investigator
Locations (2):
- United States (2):
  - University of Alabama- Birmingham, Birmingham, Alabama
  - Rick Hecht, San Francisco, California